CLINICAL TRIAL: NCT04952285
Title: The Efficacy and Safety of the Loading Dose of Tranexamic Acid in Scoliosis Surgery During Perioperative
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0215
Record Dates: First submitted 2021-06-27; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Tranexamic Acid
Keywords: tranexamic acid; Blood conservation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal saline（I）: Intravenous infusion of 0.9% saline when start to cut the skin，do not intravenous tranexamic acid during the surgery
- Tranexamic acid（II）: Intravenous infusion of tranexamic acid 1g when start to cut the skin in 1 hour

SUMMARY:
This study intends to make full use of the advantage of spinal orthopedic surgery in our medical center.Analyze the blood loss and blood coagulation function and the influence of safety of load dose tranexamic acid (TXA) in scoliosis surgery during perioperative.

ELIGIBILITY:
Inclusion Criteria:

* age:18-60 years old
* American Society of Anesthesiologists (ASA):I-II
* The spinal orthopedic undergoing elective surgery

Exclusion Criteria:

* Severe cardiopulmonary dysfunction
* Blood coagulation dysfunction
* Disorders of liver and kidney function
* Tranexamic acid allergies
* The history of pulmonary embolism and venous thrombosis of lower limbs
* Anticoagulant drugs and nonsteroidal anti-inflammatory drugs in 7 days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: age:18-60 years old；American Society of Anesthesiologists (ASA):I-II；The spinal orthopedic undergoing elective surgery
Sampling Method: Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Intraoperative blood loss | At the end of the surgery
  Intraoperative blood loss
Incision drainage Incision drainage Incision drainage after surgery | 24 hours after surgery
  Incision drainage after surgery

SECONDARY OUTCOMES:
Autologous blood doping | At the end of the surgery
  Recycle the blood during the intraoperative , back to the patient
red blood cell transfusion | At the end of the surgery
  red blood cell transfusion
Plasma infusion | At the end of the surgery
  Plasma infusion
HB | Within 1 week before surgery；1 day after surgery
  hemoglobin
WBC | Within 1 week before surgery；1 day after surgery
  White blood cells
PTL | Within 1 week before surgery；1 day after surgery
  platelet
PT | Within 1 week before surgery；1 day after surgery
  Prothrombin time
APTT | Within 1 week before surgery；1 day after surgery
  activated partial thromboplastin time
INR | Within 1 week before surgery；1 day after surgery
  International Normalized Ratio

IPD SHARING:
Plan to Share IPD: Undecided